CLINICAL TRIAL: NCT03701919
Title: Botulinum Toxin Pyloroplasty to Reduce Postoperative Nausea and Vomiting After Sleeve Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Jessica Zaman, Assistant Professor of Surgery, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5090
Record Dates: First submitted 2018-10-01; First posted 2018-10-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Bariatric Surgery; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin pyloroplasty (Experimental): Intraoperative laparoscopic intramuscular injection of 100units (10cc) of Botulinum toxin into the pylorus
  Interventions: Drug: Botulinum toxin pyloroplasty
- Normal saline pyloric injection (Placebo Comparator): Intraoperative laparoscopic intramuscular injection of 10cc normal saline into the pylorus
  Interventions: Drug: Normal saline pyloric injection

INTERVENTIONS:
Drug: Botulinum toxin pyloroplasty — Intraoperative laparoscopic injection of Botulinum toxin into the pylorus immediately following sleeve gastrectomy
  Other Names: Botox pyloropasty; Botulinum toxin A pyloroplasty
  Arms: Botulinum toxin pyloroplasty
Drug: Normal saline pyloric injection — Intraoperative laparoscopic injection of normal saline into the pylorus immediately following sleeve gastrectomy
  Arms: Normal saline pyloric injection

SUMMARY:
A common problem following sleeve gastrectomy surgery is called postoperative nausea and vomiting (PONV). This problem is uncomfortable for patients, and can also lead to other complications, including pneumonia. It is unclear what exactly causes this problem, but it may be partly caused by slow emptying of the stomach. The current treatments for PONV include medications, but these may only treat the symptoms. Botulinum toxin (BTX, brand name Botox®), produced naturally by the bacterium Clostridium botulinum and adapted for medical use, is an neurotransmitter inhibitor of the neuromuscular junction, and produces temporary muscular paralysis. BTX is widely used in cosmetic and other medical applications. Injecting BTX into the pylorus, which is the circular sphincter muscle at the end of the stomach, temporarily paralyzes the muscle, leaving it wide open, and allowing stomach contents to flow through. This effect lasts for several weeks, and then goes away. This may help prevent PONV.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) remains a common complaint after bariatric surgery such as the sleeve gastrectomy, where the prevalence is estimated to be as high as 60-80%. PONV is frequently of greater concern to patients than postoperative pain, decreasing patient satisfaction and the perioperative experience. In addition, PONV increases the risk for aspiration, dehydration, electrolyte abnormalities, incisional dehiscence, esophageal injury, and other adverse events. Finally, PONV delays postoperative diet resumption and increases hospital length of stay. Numerous medication regimens have been tried to reduce PONV after sleeve gastrectomy, with varying success. A procedure called Botulinum toxin pyloroplasty (BP), which involves injection of botulinum toxin into the muscular sphincter at the end of the stomach, called the pylorus, has been demonstrated to improve gastric emptying. The investigators hypothesize that intraoperative BP during sleeve gastrectomy will decrease rates of PONV.

Botulinum toxin type A (Botox®), produced naturally by the bacterium Clostridium botulinum and adapted for medical use, is an inhibitor of the neurotransmitter acetylcholine at the neuromuscular junction, producing flaccid muscular paralysis. The effects of Botox® injection are temporary and reversible, and its duration of action ranges from weeks to months. Botox® injection has been widely used in many contexts, most familiarly during office-based cosmetic procedures and also in disorders such as torticollis, spasticity, hyperhidrosis, bladder overreactivity, and dystonias. It has been used endoscopically to relieve achalasia and dysphagia by injection into the lower esophageal sphincter. Gastroenterologists have reported successful treatment of gastroparesis using BP, by relieving the tonic contraction of the pylorus and increasing gastric transit time. Postoperative endoscopic BP has been utilized to improve gastroparesis following gastrectomy. The use of BP during bariatric surgery has not been reported. This proposal represents the first study to evaluate the use of intraoperative BP to decrease PONV after sleeve gastrectomy.

This technique involves pyloroplasty following completion of the robot-assisted laparoscopic sleeve gastrectomy. The investigators mix 100 units of Botox® powder in 10ml of saline. Using the robot, the investigators inject the pylorus laparoscopically using an 18-gauge, 0.5-inch laparoscopic needle. Meanwhile, an assistant surgeon intubates the stomach with an endoscope, which the investigators use to assess the gastric staple line and perform a leak test. Prior to injection of Botox® into the pylorus, the investigators confirm endoscopically that the tip of the needle is not intraluminal. After first aspirating to ensure the needle is intramuscular and free from any vascular structures, the investigators then inject the pylorus with approximately 5ml of Botox®. Proper placement of the injection is confirmed by visualizing a rising weal. The anterior, superior, and inferior aspects of the pylorus are injected with approximately 5-6 injections of 1ml each. The posterior aspect of the pylorus is not injected, since this is not readily accessible from a laparoscopic approach, and also contains the major vascular structure of the pylorus, the gastroduodenal artery.

This technique has been performed at Albany Medical Center institution more than 200 times over the past four years. The Albany Medical Center Bariatric Center as participated in the Metabolic and Bariatric Surgery Accreditation for 10 years, and so has collected comprehensive and granular data on complication rates and surgical outcomes. Analysis of this data demonstrates that enteric use of Botox® is safe.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing elective sleeve gastrectomy

Exclusion criteria:

* Prior gastric surgery resulting in altered anatomy
* Documented history of postoperative nausea or vomiting
* Allergy to any of the medications used in the study
* Any use of Botulinum toxin products within six months prior to study enrollment, or plans to use Botulinum toxin products during study enrollment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Use of rescue antiemetics | During inpatient hospitalization only, an average of 2-3 days
  We will sum the number of "as needed" doses of intravenous antiemetics required by patients in both the treatment arm and the control arm of the study

SECONDARY OUTCOMES:
Patient satisfaction survey | 2 weeks postoperative
  Likert scales describing overall satisfaction with postoperative course
Subjective experience of nausea | 2 weeks postoperative
  Likert score rating subjective experience of nausea
Number of episodes of vomiting | 2 weeks postoperative
  Number of episodes of emesis
30 day readmission rate | 30 days postoperative
  30 day readmission rate
Hospital length of stay | During inpatient hospitalization only, an average of 2-3 days
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Zaman, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No